CLINICAL TRIAL: NCT05380713
Title: Surgery for Mesothelioma After Radiation Therapy Using Exquisite Systemic Therapy
Brief Title: ......SMARTEST Trial......
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-6216
Record Dates: First submitted 2022-04-08; First posted 2022-05-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Mesothelioma, Malignant
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cyclophosphamide; tremelimumab; durvalumab

STUDY DESIGN:
Intervention Model Description: This is a phase II non-blinded randomized trial designed to evaluate the benefit of low dose cyclophosphamide in sequential combination with sub-ablative radiation (Arm A) versus sub-ablative radiation alone (Arm B) before surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Radiation+Drug (Arm A) (Experimental): sub-ablative radiation plus low dose cyclophosphamide followed by surgery and adjuvant immunotherapy
  Interventions: Drug: Cyclophosphamide; Drug: Tremelimumab; Drug: Durvalumab
- Radiation alone (Arm B) (Experimental): sub-ablative radiation alone followed by surgery and adjuvant immunotherapy
  Interventions: Drug: Tremelimumab; Drug: Durvalumab

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide will be applied in the neoadjuvant setting
  Arms: Radiation+Drug (Arm A)
Drug: Tremelimumab — tremelimumab-durvalumab in adjuvant setting
Drug: Durvalumab — tremelimumab-durvalumab in adjuvant setting

SUMMARY:
The SMARTEST trial is a phase II non-blinded randomized trial designed to evaluate the benefit of low dose cyclophosphamide in sequential combination with sub-ablative radiation (Arm A) versus sub-ablative radiation alone (Arm B) before surgery as well as the safety and efficacy of consolidation tremelimumab-durvalumab for eligible patients after surgery in both arms.

DETAILED DESCRIPTION:
This study has two parts. In the first part of the study the investigators are exploring the benefit of using low dose Cyclophosphamide in combination with low dose radiation before surgery and in the second part of the study the investigators are exploring safety and efficacy of using a combination of immunotherapy drugs, tremelimumab-durvalumab, after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Age ≥ 18 years at the time of study entry
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Body weight >30 kg
5. Adequate normal organ and marrow function as defined below:
6. Haemoglobin ≥9.0 g/dL
7. Absolute neutrophil count (ANC ≥1.0 × 109 /L)
8. Platelet count ≥75 × 109/L
9. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
10. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
11. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

    Males:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

    Females:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
13. Must have a life expectancy of at least 12 weeks
14. Tumor amenable to biopsy
15. Histologically proven mesothelioma
16. Previously untreated mesothelioma
17. Stage I to III according to the 8th edition of the TNM staging system based on CT chest-abdomen and fluorodeoxyglucose (FDG) PET scan. Tumor assessment by CT and PET scan must be performed within 60 days prior to randomization.
18. Suitable for surgery and combined modality therapy in the opinion of the investigator

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 8 weeks
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
3. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy (including radiation , surgery and low dose cyclophosphamide) with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
4. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
5. Previous thoracic irradiation
6. Serious non-malignant disease (cardiovascular, pulmonary, systemic lupus erythematosus, scleroderma) that would preclude definitive radiation therapy
7. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
8. History of allogenic organ transplantation.
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   5. Patients with celiac disease controlled by diet alone
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
11. Patients with a history of other malignancies, except non-active malignancy that does not require treatment, nor anticipated to require treatment for the duration of the study, and in the opinion of the investigator would not pose a risk of increased toxicity, or difficulty to follow the protocol and assess endpoints of the study
12. History of leptomeningeal carcinomatosis
13. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry.
14. Distant metastatic disease (M1), including brain metastasis or spinal cord compression
15. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
16. History of active primary immunodeficiency
17. Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Adjust wording as necessary and consider evaluating at screening for studies with known hepatotoxicity or other relevant requirements.
18. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
19. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
    4. Use of immunosuppressive medications for the management of IP-related AEs
    5. Use in patients with contrast allergies
    6. A temporary period of steroids will be allowed if clinically indicated and considered to be essential for the management of non-immunotherapy related events experienced by the patient (e.g., chronic obstructive pulmonary disease, radiation, nausea, etc.)
20. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
21. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or180 days after the last dose of durvalumab and tremelimumab combination therapy.
22. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
23. Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
24. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.
25. Failure to provide consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
CD8 TILs density / gross tumor volume (GTV) | Up to five years
  The primary objective of the study is to demonstrate that low dose cyclophosphamide in combination with sub-ablative radiation can enhance the anti-tumoral immune response compared to sub-ablative radiation alone

SECONDARY OUTCOMES:
Survival | Up to five years
  Demonstrate the safety and efficacy of tremelimumab-durvalumab in the adjuvant setting after sub-ablative radiation and surgery with and without low dose cyclophosphamide

OTHER OUTCOMES:
Proportional change in circulating CD8 RA+ effector memory T cells, Proportional change in circulating CD4 RA+ effector memory T cells | Up to five years
  Identify biomarkers associated with prognosis and response to therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided